CLINICAL TRIAL: NCT02481986
Title: Asthma Action at Erie Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Erie Family Health Center (Other Government); Rush University Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Molly A. Martin, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-0026; R01HL123797 (NIH)
Record Dates: First submitted 2015-06-05; First posted 2015-06-25 (Estimated); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma; Children
MeSH Terms: conditions — Asthma | interventions — Community Health Workers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Community health worker (Experimental): Participants in this arm will be offered 10 home visits in a 12-month period from community health workers (CHWs). Visits will cover a core asthma curriculum and provide social support.
  Interventions: Behavioral: Community Health Worker
- Certified asthma educator (Active Comparator): Participants in this arm will be offered 2 education sessions with a certified asthma educator in the clinic at start of the study and again at 6-months. These sessions will be followed by a telephone call from the certified asthma educator several weeks after the sessions.
  Interventions: Behavioral: Certified asthma educator

INTERVENTIONS:
Behavioral: Community Health Worker — A community health worker is para-professional who performs education, case management, and social support.
  Arms: Community health worker
Behavioral: Certified asthma educator — A certified asthma educator has is certified and performs asthma education.
  Arms: Certified asthma educator

SUMMARY:
The Asthma Action at Erie Trial compares the current best practice in asthma self-management education (certified asthma educator services) to an integrated community health worker (CHW) home intervention in which the real-life challenges of patients and the health care system are taken fully into account. This trial will provide clarity as to the expected effect size, cost savings, and resources needed to integrate asthma CHWs into clinical practice.

DETAILED DESCRIPTION:
The Asthma Action at Erie Trial will test the ability of a community health worker (CHW) intervention with three important modifications to achieve asthma control in high-risk children. These modifications are: 1) CHWs will be integrated into both the clinical and the home setting, 2) A system for directly addressing mental health and psychosocial barriers will be provided, and 3) Participants will be provided only materials and equipment for trigger remediation that are supported by the current medical reimbursement system. To test this intervention, a two-arm behavioral randomized controlled trial (N=220) will be conducted in partnership with a federally-qualified health center (FQHC) serving a low income, minority population that is at high-risk for significant asthma morbidity. The intervention arm will receive an integrated CHW home intervention for pediatric asthma education. The comparison arm will received clinic-based certified asthma educator (AE-C) services. Primary Aim 1 is to assess the efficacy of the integrated CHW home asthma intervention, relative to clinic-based AE-C education over 12-months, as demonstrated by asthma control. Specific Aim 2 is to assess maintenance of intervention efficacy, as demonstrated by asthma control at 18 and 24 months after randomization. Specific Aim 3 is to determine the cost-effectiveness at 12-months of CHW and AE-C intervention delivery, and additional costs or savings related to asthma exacerbations at 12- and 24-months. Specific Aim 4 is to assess the efficacy of the integrated CHW home asthma intervention relative to clinic-based AE-C education, as demonstrated by asthma control, among those experiencing depression, stress, and/or a post-traumatic stress disorder.

ELIGIBILITY:
Inclusion Criteria:

* Child is a patient at Erie Family Health Center
* Child is age 5-16 at the start of the study
* Child lives with the index caregiver at least 5 days out of the week
* Child has uncontrolled asthma. This is defined as a score of 1.25 or greater on the Asthma Control Questionnaire, or report of oral corticosteroid use in the past year
* Family has a working telephone

Exclusion Criteria:

* Exclusion criteria include family not fluent in English or Spanish, family lives in temporary housing such as a shelter, caregiver does not have permanent custody of child, or child has significant developmental delays or co-morbidities that would limit their ability to participate in the program.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 223 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Erie Family Health Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Lalji R, Koh L, Francis A, Khalid R, Guha C, Johnson DW, Wong G. Patient navigator programmes for children and adolescents with chronic diseases. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD014688. doi: 10.1002/14651858.CD014688.pub2. PMID 39382077
- [Derived] Weinstein SM, Pugach O, Rosales G, Mosnaim GS, Orozco K, Pappalardo AA, Martin MA. Psychosocial Moderators and Outcomes of a Randomized Effectiveness Trial for Child Asthma. J Pediatr Psychol. 2021 Jul 20;46(6):673-687. doi: 10.1093/jpepsy/jsab011. PMID 33616185
- [Derived] Weinstein SM, Pugach O, Rosales G, Mosnaim GS, Walton SM, Martin MA. Family Chaos and Asthma Control. Pediatrics. 2019 Aug;144(2):e20182758. doi: 10.1542/peds.2018-2758. Epub 2019 Jul 9. PMID 31289192
- [Derived] Mosnaim GS, Weinstein SM, Pugach O, Rosales G, Roy A, Walton S, Martin MA. Design and baseline characteristics of a low-income urban cohort of children with asthma: The Asthma Action at Erie Trial. Contemp Clin Trials. 2019 Apr;79:55-65. doi: 10.1016/j.cct.2019.02.006. Epub 2019 Feb 14. PMID 30772471

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Community Health Worker | Certified Asthma Educator
Started | 108 | 115
Completed | 103 | 106
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Community Health Worker | Certified Asthma Educator | Total
Number analyzed (Participants) | 108 | 115 | 223
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 108 | 115 | 223
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (2.9) | 9.5 (3.2) | 9.4 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 52 | 98
  Male | 62 | 63 | 125
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One family did not answer child race. Note that race and ethnicity were asked as separate questions.
  Participants
    Hispanic ethnicity child | 92 | 98 | 190
    Not Hispanic ethnicity child | 16 | 17 | 33
    Black race child: number analyzed (Participants) | 108 | 114 | 222
    Black race child | 18 | 21 | 39
    Not Black race child: number analyzed (Participants) | 108 | 114 | 222
    Not Black race child | 90 | 93 | 183
Region of Enrollment [Number; unit: participants]
  United States | 108 | 115 | 223

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Test/Childhood Asthma Control Test at 12-months
Description: Asthma Control Test (12 years or older) or Childhood Asthma Control Test (under 12 years old) minimum 5, maximum 27, higher score means better asthma control
Time Frame: assessed 12-months from baseline, assessed over past 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Community Health Worker | Certified Asthma Educator
Number analyzed (Participants) | 103 | 106
score on a scale | 21.23 [19.82 to 22.63] | 20.58 [19.31 to 21.85]

2. Primary Outcome: Activity Limitation at 12-months
Description: Days of activity limitation over past 14 days minimum 0, maximum 14, higher means worse asthma control
Time Frame: assessed 12-months after baseline, assessed over past 14 days
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio of days
Arm/Group | Community Health Worker | Certified Asthma Educator
Number analyzed (Participants) | 103 | 106
ratio of days | 0.42 [0.04 to 0.80] | 0.88 [0.52 to 1.23]

3. Secondary Outcome: Asthma Control Questionnaire at 12-months
Description: Asthma Control Questionnaire minimum 0, maximum 6, higher score means worse asthma control
Time Frame: assessed 12-months after baseline, prior week assessed
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Community Health Worker | Certified Asthma Educator
Number analyzed (Participants) | 103 | 106
score on a scale | 0.80 [0.57 to 1.04] | 0.88 [0.66 to 1.09]

4. Secondary Outcome: Health Care Utilization at 12-months
Description: Any ED visits or hospitalizations for asthma (each ED visit or hospitalization is a single event, ED visits that transition into hospitalizations are coded as one event)
Time Frame: assessed 12-months after baseline, assessed from baseline to 12-months
Measure: Least Squares Mean (95% Confidence Interval); unit: events
Arm/Group | Community Health Worker | Certified Asthma Educator
Number analyzed (Participants) | 103 | 106
events | 0.11 [0.07 to 0.18] | 0.20 [0.13 to 0.28]

5. Secondary Outcome: Costs of Intervention Delivery
Description: This measure is the total dollars spent to deliver the intervention by arm. Costs include CHW and AE-C salaries, supervision, training costs, and intervention materials that resulted in 84 AE-visits and 722 CHW visits.
Time Frame: assessed 12-months from baseline, assessed from baseline to 12-months
Measure: Number; unit: dollars spent per arm on intervention
Arm/Group | Community Health Worker | Certified Asthma Educator
Number analyzed (Participants) | 108 | 115
dollars spent per arm on intervention | 53390 | 11373

ADVERSE EVENTS:
Time Frame: 24 months per participant
Arm/Group | Community Health Worker | Certified Asthma Educator
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/115
Other Adverse Events (participants affected / at risk) | 0/108 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT02481986/Prot_SAP_000.pdf